CLINICAL TRIAL: NCT07276815
Title: Gathering of Results in Eligible Asian Obese Populations About Safety and Effectiveness of Overstitch ESG Trial
Brief Title: OverStitch NXT Endoscopic Suture System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E7241
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Roll-in Cases (Other): ESG combined with lifestyle management for 12 months
  Interventions: Device: OverStitch NXT Endoscopic Suture System
- Treatment group (Experimental): ESG combined with lifestyle management for 12 months.
  Interventions: Device: OverStitch NXT Endoscopic Suture System
- Control group (No Intervention): Lifestyle management alone for 12 months, followed by evaluation. Eligible participants may undergo ESG afterward.

INTERVENTIONS:
Device: OverStitch NXT Endoscopic Suture System — The OverStitch NXT Endoscopic Suture System is indicated for the endoscopic placement of anchor-sutures. Anchor sutures can be placed for endoscopic sleeve gastroplasty（ESG）.
  Arms: Roll-in Cases; Treatment group

SUMMARY:
To demonstrate the safety and efficacy of OverStitch NXT Endoscopic Suture System for endoscopic sleeve gastroplasty（ESG） in obese populations to support the registration of OverStitch NXT for ESG indication.

DETAILED DESCRIPTION:
The study is a prospective, multicenter, randomized controlled trial

This study is planned to be conducted at 10 sites, with each center initially enrolling 2 roll-in cases (totaling 20 cases). After each site completes the enrollment of its roll-in cases, the remaining subjects will be randomly divided into two groups (the treatment group and the control group) via a central randomization system. Each group will ultimately enroll 58 subjects, resulting in a total sample size of 136 for the study.

Roll-in Cases: ESG combined with lifestyle management for 12 months. treatment group: ESG combined with lifestyle management for 12 months. control group: Lifestyle management alone for 12 months, followed by evaluation. Eligible participants may undergo ESG afterward.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, or subjects who have reached the legal age for signing informed consent in accordance with local laws and regulations.
2. BMI ≥ 32.5 kg/m²; or BMI ≥ 27.5 kg/m² combined with type 2 diabetes mellitus (regardless of the effectiveness of medical treatment for type 2 diabetes); or BMI between 27.5 kg/m² and 32.5 kg/m² with ineffective medical weight loss or combined with other obesity-related diseases for which medical treatment is ineffective.
3. Willing to comply with the long-term strict dietary restrictions required by the surgery.
4. Capable of providing informed consent, able to complete all routine follow-up visits, and willing to abide by the protocol requirements, including signing the informed consent form, completing relevant examinations, and receiving dietary counseling.
5. Females of childbearing potential (i.e., premenopausal or not sterilized) must agree to use adequate contraceptive measures.

Exclusion Criteria:

1. History of foregut or gastrointestinal (GI) surgery (except uncomplicated cholecystectomy or appendectomy)
2. Prior gastrointestinal surgery with sequelae, i.e. obstruction, and/or adhesive peritonitis or known abdominal adhesions.
3. Prior open or laparoscopic bariatric surgery.
4. Prior surgery of any kind on the esophagus or any type of hiatal hernia surgery.
5. Any inflammatory disease of the gastrointestinal tract including severe (LA Grade C or D) esophagitis, gastric ulceration, duodenal ulceration, specific inflammation such as Crohn's disease, and the doctor judges that it may affect the operation or efficacy of ESG.
6. Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresia or stenosis.
7. History of gastrointestinal stromal tumors, gastrointestinal cancer, low-grade or high-grade gastric intraepithelial neoplasia, or familial or non-familial adenomatous polyposis syndrome.
8. Gastric masses or untreated gastric polyps with a diameter > 1 cm.
9. Hiatal hernia (Z-line displacement above the diaphragm > 4 cm) or severe/refractory gastroesophageal reflux symptoms, which the physician judges may affect the performance or prognosis of ESG.
10. Structural abnormalities of the esophagus or pharynx that may impede endoscopic passage (e.g., strictures or diverticula), which the physician judges may affect the performance or prognosis of ESG.
11. Gastrointestinal motility disorders (e.g., achalasia, severe esophageal motility disorders, gastroparesis, or intractable constipation), which the physician judges may affect the performance or prognosis of ESG.
12. Evidence of untreated psychiatric or eating disorders, such as major depression, schizophrenia, substance abuse, binge eating disorder, or bulimia nervosa.
13. Coagulopathy with INR > 1.5 that cannot be corrected (per physician's judgment) or requirement for continuous full anticoagulant therapy, and/or any underlying diseases associated with high bleeding risk.
14. Insulin-dependent diabetes mellitus (type 1 or type 2), or high likelihood of requiring insulin therapy within the next 12 months.
15. Decompensated cirrhosis, or acute/chronic liver dysfunction that the physician judges make the subject unsuitable for ESG treatment.
16. Diagnosis of autoimmune connective tissue diseases (e.g., systemic lupus erythematosus, scleroderma) or immunocompromise, which the physician assesses may affect the performance or prognosis of ESG.
17. Known history of endocrine diseases affecting body weight (e.g., Cushing's syndrome, uncontrolled hypothyroidism, or hyperthyroidism), which the physician assesses may affect the performance or prognosis of ESG.
18. Anemia: Hemoglobin (Hgb) < 110 g/L for females; Hgb < 120 g/L for males.
19. Any other medical conditions precluding elective endoscopy, such as poor general health, history of severe renal, hepatic, cardiac, and/or pulmonary diseases, and/or severe or uncontrolled psychiatric illnesses or abnormalities that may impair the patient's ability to understand or comply with follow-up visits and lifestyle interventions.
20. Active psychological issues as determined by a psychologist or psychiatrist, precluding participation in lifestyle modification programs.
21. Unwillingness to participate in the established medically supervised dietary and behavioral modification programs, as well as routine medical follow-up.
22. Daily treatment with prescribed high-dose aspirin (> 80 mg per day), non-steroidal anti-inflammatory drugs (NSAIDs), antiplatelet agents, anticoagulants, corticosteroids, immunosuppressants, or other gastric irritant medications.
23. Interval use of medications that may be affected by changes in gastric emptying (e.g., antiepileptic drugs or antiarrhythmic drugs).
24. Inability or unwillingness to take prescribed proton pump inhibitor (PPI) medications.
25. Current use of weight loss medications or other weight loss devices or use within the past 90 days.
26. Current participation in a clinical trial involving investigational drugs or devices, or participation in such a trial within 30 days prior to enrollment in this study.
27. Use of intragastric devices within 30 days prior to this study, which the physician assesses may affect the performance or prognosis of ESG.
28. Unwillingness to avoid any reconstructive and/or plastic surgeries that may affect body weight during the study (e.g., mammoplasty, liposuction).
29. Other conditions deemed unsuitable for endoscopy or ESG treatment by the investigator, including but not limited to conditions that the investigator believes may expose the subject to significant risks, confound study results, increase risks associated with endoscopy and/or endoscopic procedures, or substantially interfere with the subject's participation in the study.
30. Pregnancy, lactation, or intention to become pregnant during the study (for females of childbearing potential).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2026-07-31 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
%TBWL (Defined as the percentage of total body weight loss) | At 12 months after the intervention.
  %TBWL is defined as the percentage of total body weight loss
The response rate at the 12th month after the intervention | At 12 months after the intervention
  Response is defined as having a percentage of total body weight loss (%TBWL) of ≥ 5%